CLINICAL TRIAL: NCT03691519
Title: Prevention of Cognitive Decline in Older Adults With Low Dha/Epa Index in Red Blood Cells
Acronym: LO-MAPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RC31/16/8752; 2016-A01450-51 (Other: ID-RCB)
Record Dates: First submitted 2018-06-14; First posted 2018-10-01 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Alzheimer Disease
Keywords: Low OMega 3; Preventive trial; low RBC DHA/EPA index
MeSH Terms: conditions — Alzheimer Disease | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned in a 1:1 ratio to one of the following 2 groups: (i) DHA+EPA supplement or (ii) placebo. A computer-generated randomisation procedure will be used with stratification by centre. A centralised Interactive Voice Response System will be used to identify which group to allocate and which lot number to administrate
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study will be a double-blind trial. The packaging, presentation, and labelling of products will ensure the blinding of both the medical team and the patient. The treatment arms in this study will be differentiated only by treatment numbers. Treatment arms will be allocated treatment numbers according to the previously established randomisation table.
  Neither the investigating doctors nor the patients will be aware of the treatment arm to which the patients have been allocated until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): During the 18 months placebo-controlled period, participants will ask to consume 3 identical 1g vegetarian control capsules (containing a 1:1 ratio of corn oil and soy oil) per day. During the following 18-month open-label extension period, placebo subjects are switched to active treatment.
  36 months consisting of a 18-month placebo-controlled period followed by a 18-month open-label extension period wherein all participants will receive active treatment
  Interventions: Dietary Supplement: Placebo
- Omega-3 treatment (Experimental): During the entire length of the study (that is, both the placebo-controlled and open-label extension periods), participants in the intervention (Omega-3 treatment) arm will ask to consume 3- 1g softgel vegetarian capsules of DHA-O per day as a single dose for 36 months; each 1g capsule of DHA-0 providing 324 mg DHA and 185 mg EPA (total daily DHA+EPA dose = 1.53 g/day).
  Interventions: Drug: Omega-3 treatment

INTERVENTIONS:
Drug: Omega-3 treatment — Patient in the "treatment comparative arm will consume 3- 1g softgel vegetarian capsules of DHA-O per day as a single dose for 36 months; each 1g capsule of DHA-0 providing 324 mg DHA and 185 mg EPA (total daily DHA+EPA dose = 1.53 g/day).
  Other Names: Dietary intervention
  Arms: Omega-3 treatment
Dietary Supplement: Placebo — The appearance and taste of the placebo will be similar to those of the active ingredient. Placebo capsules contained a 1:1 ratio of corn oil and soy oil.
  36 months consisting of a 18-month placebo-controlled period followed by a 18-month open-label extension period wherein all participants will receive active treatment. Active treatment consists of 1.53 g /day dose of DHA-0 (972 mg /day DHA + 555 mg /day EPA; 3 caps /day).
  For the 18 months placebo-controlled period (n=200/arm): 1.53 g /day dose of DHA-0 (972 mg /day DHA + 555 mg /day EPA; 3 caps /day) or placebo (3 similar pills /day).
  Arms: Placebo

SUMMARY:
LO MAPT is an 18-month, phase III, multicenter, randomized, placebo-controlled, 2 parallel groups trial, followed by a 18-month open-label extension phase, to evaluate the efficacy of omega-3 supplementation on cognitive decline in older adults with low DHA/EPA status and subjective memory complaints or family history of Alzheimer disease.

DETAILED DESCRIPTION:
LO-MAPT will also assess the effect of an audiovisual aid, compared with traditional paper participant information sheet only, on participants' understanding of the protocol, as well as on drop-out, adherence and clinical outcome in older adults at risk of cognitive decline. In addition to the main LO-MAPT study procedures, in two centers, half of the subjects will receive an audiovisual aid in addition to the standard information sheet.

The primary objective of LO MAPT is to demonstrate the efficacy of a 18-month intervention with a supplementation of omega-3 (DHA+EPA) on cognitive decline as measured by a composite score of neuropsychological assessments in older adults with low DHA/EPA status (RBC DHA/EPA index ≤ 4.83%) and subjective memory complaints or family history of Alzheimer's disease.

Subjects will be randomly assigned in a 1:1 ratio to one of the following 2 groups: (i) DHA+EPA supplement or (ii) placebo. A computer-generated randomisation procedure will be used with stratification by centre. A centralised Interactive Voice Response System will be used to identify which group to allocate and which lot number to administer. A document describing the randomization procedure will be kept confidentially by the Methodology and Data Management Centre. All participants and study staff will be blinded to DHA+EPA supplement/placebo assignment: all participants will receive soft capsules of exactly the same appearance and taste.

ELIGIBILITY:
Inclusion Criteria:

* RBC DHA/EPA index ≤ 4.83% with at least one of the following criteria:
* subjective memory complaint,
* family history of Alzheimer's disease;
* Mini-Mental State Examination (MMSE) score ≥ 24;
* Have a study partner that is willing to participate as a source of information and has at least weekly contact with the participant (contact can be in person, via telephone or electronic communication);
* Sufficient vision and hearing to complete study protocol procedures based on medical judgment;
* Have general health status that will not interfere with the ability to complete the study;
* Willing and able to participate and to give written consent to comply with study procedures;
* Covered by a health insurance system.

Exclusion Criteria:

* Criteria related to diseases:
* Known presence of dementia or Alzheimer's disease (DSMIV criteria);
* Dependency for basic activities of daily living (ADL score <4);
* Presence of serious diseases, which could be life-threatening in the short term.
* Criteria related to treatments:
* Taking of supplements containing omega-3 (apart from food) within the past 6 months and/or taking omega-3 at inclusion.
* Criteria related to subjects:
* Visual or hearing impairments incompatible with performance and/or interpretation of the neuropsychological tests;
* History or presence of any previous condition (severe depression or generalized anxiety) that could, in the opinion of the investigator, interfere with the results of the study or expose the subject to an additional risk;
* Subjects deprived of their liberty by administrative or judicial decision, or under guardianship or admitted to a healthcare or social institution (subjects in non-assisted living facilities could be recruited);
* Participation in another clinical study in the previous month or participation scheduled during the study;
* Food allergy.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 774 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of Composite Z-score which evaluate cognitive performance | 18 months
  This composite score will be built of Z-scores of these components. As this criterion will be assessed during each visit (the enrolment visit and the 4 follow-up visits), the analysis will be carried out by taking repeat measurements, taking the correlated of the data into consideration, evaluating Change from Baseline

SECONDARY OUTCOMES:
FCSRT Test | 18 months
  Tests included in the composite score will be analyzed independently The Free and Cued Selective Reminding test (FCSRT) is a memory test that controls attention and acquisition : Verbal learning with 16-word free and indexed recall test. Each word is identified by a semantic category. Word encoding is controlled. The total learning score is equal to the sum of the free and indexed recall. The maximum score is 48.
MMSE total score | 18 months
  MMSE (MINI MENTAL STATE EXAMINATION) total score : 30-question general cognitive function assessment. The maximum score is 30.
Category Naming Test (CNT) | 18 months
  The CNT is a semantic verbal fluency test which assesses spontaneous production of words belonging to the same category within a certain time (i.e. the animal category).

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Vellas, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No